CLINICAL TRIAL: NCT05040334
Title: Role of Prophylactic Antibiotics in Preventing Pelvic Infection After Surgical Evacuation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Mohamed Mahmoud Eid, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Cairo University Obygyn
Record Dates: First submitted 2021-08-14; First posted 2021-09-10 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Antibiotics Causing Adverse Effects in Therapeutic Use

STUDY DESIGN:
Intervention Model Description: Group 1;receiving antibiotic prophylaxis Group 2; Not receiving antibiotics
Who Masked: Participant
Masking Description: 138 identical envelops, half of them filled with a label(Group 1) who are the "Prophylactic antibiotic" group with all instruction details, while the other half are labelled (group 2) who are the "Placebo" group with all instruction details. All envelops will be prepared by the investigator and sealed before starting enrollment. After enrollment, each participant will be allowed to choose one envelop to determine to which group she will be assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group(1) (Active Comparator): 69 patients receiving a single dose of oral doxycycline (200 mg) and metronidazole (500 mg)tablets
  Interventions: Drug: Group 1: Antibiotic receiving group
- Group (2) (Placebo Comparator): 69 patients receiving placebo
  Interventions: Drug: Group 1: Antibiotic receiving group

INTERVENTIONS:
Drug: Group 1: Antibiotic receiving group — Group 1; receiving antibiotic prophylaxis; single dose of oral doxycycline (200 mg) tablet and metronidazole (500 mg) tablet 2 hours before the surgical evacuation Group B ;receiving placebo 2 hours before the surgical evacuation
  Other Names: Group 2 :placebo receiving group

SUMMARY:
To determine the role of antibiotic prophylaxis in the surgical management of miscarriage.

DETAILED DESCRIPTION:
Patients will be randomized to receive either prophylactic antibiotic [a single dose of oral doxycycline (200 mg) and metronidazole (500 mg)] or placebo using identical sealed envelopes.Included cases are those with early miscarriage (within the first trimester 12 6/7 weeks of gestation) , missed or incomplete miscarriage, undergoing surgical management will be included in the study.

Technique:

The investigators will prepare 138 identical envelops, half of them filled with a label group(1) who are the group to receive the antibiotic prophylaxis with all instruction details, while the other half filled with a label identifying ( group 2) who are the placebo group. All envelops will be prepared by the investigator and sealed before starting enrollment. After enrollment, each participant will be allowed to choose one envelop to determine to which group the patient will be assigned to.

ELIGIBILITY:
Inclusion criteria:

* Maternal age :18-35 years
* Gestational age: up to 12 6/7 weeks of gestation (confirmed by a reliable date for the last menstrual period or /and 1st trimester ultrasound scan).
* Singleton miscarriage
* Type of miscarriage: Incomplete or Missed miscarriage
* Surgical evacuation will be done within 2 weeks of diagnosis of miscarriage .

Exclusion criteria:

* Maternal age: younger than 18 years
* Induced miscarriage of pregnancy
* Septic miscarriage
* Evidence of infection
* Morbid obesity (BMI≥40kg/m2)
* Allergy to prophylactic antibiotics (i.e., doxycycline or metronidazole)
* Antibiotics use within 7 days before randomization

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 138 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Change of pelvic infection after surg ical evacuation of miscarriage with use of antibiotic prophylaxis. | 2 weeks from surgery
  White cell count >12 *10^9 cells / L by CBC

SECONDARY OUTCOMES:
Change in the risk of severe puerperal sepsis following the surgical procedure | 2 weeks from surgery
  Signs of puerperal sepsis in form of puerperal pyrexia >38 C and/or purulent vaginal discharge

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Mo Eid, Ass.prof., Study Director — Cairo University; Nihal Mo El-Demiry, lecturer, Principal Investigator — Cairo University
Locations (1):
- Department of Obstetrics and Gynecology, Kasr Al-Ainy University Hospital, Cairo University., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided